CLINICAL TRIAL: NCT01462370
Title: A Phase III, Randomized, Active-Comparator-Controlled, 2-period, Crossover, Double-Blind Study in China to Assess the Safety and Efficacy of Etoricoxib 120 mg Versus Ibuprofen up to 2400 mg (600 mg Q6h) in the Treatment of Patients With Primary Dysmenorrhea
Brief Title: Study to Assess the Safety and Efficacy of Etoricoxib Versus Ibuprofen in the Treatment of Dysmenorrhea (MK-0663-145 AM1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-145
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Etoricoxib; Ibuprofen; Acetaminophen; Saridon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etoricoxib+placebo ibuprofen then placebo etorcoxib+ibuprofen (Experimental): Participants will receive one tablet (active or placebo etoricoxib) and 3 capsules (active or placebo ibuprofen) as their first dose of study medication in Cycle 1 and Cycle 2. They can also take 3 capsules (active or placebo ibuprofen) up to 3 times more per day in Cycle 1 and Cycle 2.
  Interventions: Drug: Etoricoxib; Drug: Ibuprofen; Drug: Placebo to etoricoxib; Drug: Placebo to ibuprofen; Drug: Acetaminophen 250 mg, isopropylantipyrine 150 mg and anhydrous caffeine 50 mg
- Ibuprofen+placebo etoricoxib then etoricoxib+placebo ibuprofen (Experimental): Participants will receive one tablet (active or placebo etoricoxib) and 3 capsules (active or placebo ibuprofen) as their first dose of study medication in Cycle 1 and Cycle 2. They can also take 3 capsules (active or placebo ibuprofen) up to 3 times more per day in Cycle 1 and Cycle 2.
  Interventions: Drug: Etoricoxib; Drug: Ibuprofen; Drug: Placebo to etoricoxib; Drug: Placebo to ibuprofen; Drug: Acetaminophen 250 mg, isopropylantipyrine 150 mg and anhydrous caffeine 50 mg

INTERVENTIONS:
Drug: Etoricoxib — Etoricoxib 120 mg tablet given orally for one dose.
Drug: Ibuprofen — Ibuprofen 600 mg (three 200-mg capsules) given orally up to four times a day as needed, for a maximum of 2400 mg/day.
Drug: Placebo to etoricoxib — Placebo to etoricoxib, one tablet.
Drug: Placebo to ibuprofen — Placebo to ibuprofen, up to four 3-capsule doses.
Drug: Acetaminophen 250 mg, isopropylantipyrine 150 mg and anhydrous caffeine 50 mg — Provided to participants as rescue medication. Participants may take 2 tablets at a time and up to 3 doses within 24 hours for rescue purposes.
  Other Names: Saridon

SUMMARY:
This is a study to determine the overall analgesic effect of a single oral dose of etoricoxib compared to ibuprofen in participants with moderate-to-severe primary dysmenorrhea.

DETAILED DESCRIPTION:
Participants who meet all the study entry criteria will be randomly allocated to 2 possible sequences of the 2 treatment regimens over the course of 2 menstrual cycles.

In treatment sequence 1, participants will receive etoricoxib 120 mg daily in menstrual cycle 1, and ibuprofen up to 2400 mg/daily in menstrual cycle 2. In treatment sequence 2, participants will receive ibuprofen up to 2400 mg/daily in menstrual cycle 1 and etoricoxib 120 mg daily in menstrual cycle 2.

ELIGIBILITY:
Inclusion Criteria:

* Agree to remain abstinent or use double-barrier contraception throughout the study. Participants who are status post tubal ligation are exempt from this requirement.
* Moderate or severe primary dysmenorrhea during a minimum of 4 of the previous 6 menstrual cycles. Moderate: Over-the-counter analgesics provide significant relief in most menstrual cycles; discomfort interferes with usual activity. Severe: Over-the-counter analgesics not consistently effective, or prescription analgesics required in at least some menstrual cycles; discomfort is incapacitating causing an inability to work or do usual activity.
* Willing to limit alcohol intake to 2 drinks or equivalent per day for the duration of the study and follow-up period as well as to avoid exercise during the first 24 hours postdose in each menstrual cycle.
* Able to read, understand, and complete diary.

Exclusion Criteria:

* Use of an intrauterine device. Pregnant, breast feeding, or <6 weeks postpartum.
* Active gastric ulcer or history of inflammatory bowel disease.
* Uncontrolled hypertension.
* Uncontrolled diabetes mellitus or renal disease.
* Class II-IV congestive heart failure.
* Coronary artery bypass graft surgery, angioplasty, myocardial infarction, cerebrovascular accident or transient ischemic attack within the past 6 months.
* Unstable angina.
* Mild, moderate, or severe hepatic insufficiency.
* Any personal or family history of an inherited or acquired bleeding disorder.
* History of neoplastic disease; Exceptions: 1)adequately treated basal cell carcinoma or carcinoma in situ of the cervix; 2) other malignancies which have been successfully treated > or equal to 5 years prior to screening. Participants with a history of leukemia, lymphoma, malignant melanoma, and myeloproliferative disease are ineligible for the study regardless of the time since treatment.
* Allergic to etoricoxib, ibuprofen, acetaminophen, indomethacin, or other nonsteroidal anti-inflammatory drugs (NSAIDs), or cyclooxygenase (COX)-2 inhibitors, or to components in Saridon (propyphenazone/paracetamol/caffeine).
* Recent history of chronic analgesic or tranquilizer use or dependence.
* Morbidly obese and demonstrates significant health problems stemming from the obesity.
* Current user of recreational or illicit drugs or had a recent history of drug or alcohol abuse or dependence.
* Participated in another clinical study within the last 4 weeks.
* Not able to swallow oral medications: surgical or anatomical conditions that will preclude from swallowing and absorbing oral medications on an ongoing basis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

REFERENCES:
- [Result] Yu Q, Zhu X, Zhang X, Zhang Y, Li X, Hua Q, Chang Q, Zou Q, Di W, Yao Y, Yu W, Liu J, Mehta A, Yan L. Etoricoxib in the treatment of primary dysmenorrhea in Chinese patients: a randomized controlled trial. Curr Med Res Opin. 2014 Sep;30(9):1863-70. doi: 10.1185/03007995.2014.925437. Epub 2014 Jun 30. PMID 24960147

RESULTS

PARTICIPANT FLOW:
Groups:
- Etoricoxib 120 mg/ Ibuprofen Up to 2400 mg: Etoricoxib 120 mg tablet given orally or one dose in menstrual cycle 1. In menstrual cycle 2, ibuprofen was administered at a dose of 600 mg every 4 hours as needed up to 2400 mg/day.
- Ibuprofen Up to 2400 mg / Etoricoxib 120 mg: Ibuprofen 600 mg given orally up to for times a day as needed for a maximum of 2400 mg/day in menstrual cyle 1. In menstrual cycle 2, etoricoxib 120 mg ws given orally for one dose.
Period: Overall Study
Arm/Group | Etoricoxib 120 mg/ Ibuprofen Up to 2400 mg | Ibuprofen Up to 2400 mg / Etoricoxib 120 mg
Started | 69 | 70
Completed | 68 | 65
Not Completed | 1 | 5
Not completed — Lack of Qualifying Event | 1 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All participants randomized into the study.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 139
Age, Customized [Number; unit: Participants]
  <=20 years | 14
  21-29 years | 118
  >=30 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Pain Relief Score Over the First 6 Hours (TOPAR6) After the Initial Dose
Description: TOPAR6 was calculated by multiplying the pain relief (PR) score (0- to 4-point scale, with 0=None, and 4=Complete for pain relief) at each time point by the duration (in hours) since the preceding time point, and summing these weighted values up to 6 hours post the initial Day 1 dose. The range of TOPAR6 score is 0 to 24, with increasing scores indicating greater pain relief.
Time Frame: Baseline and 0.5, 1, 1.5, 2, 3, 4, 5 and 6 hours
Population: The population consisted of all participants that received at least one dose of study treatment and had at least one TOPAR6 observation up to 6 hours post initial dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Groups:
- Etoricoxib 120 mg: Etoricoxib 120 mg tablet given orally for one dose.
- Ibuprofen up to 2400 mg: Ibuprofen 600 mg (three 200-mg capsules) given orally up to four times a day as needed, for a maximum of 2400 mg/day.
Arm/Group | Etoricoxib 120 mg | Ibuprofen up to 2400 mg
Number analyzed (Participants) | 130 | 130
Score on a Scale | 17.38 (0.37) | 16.49 (0.37)
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Ibuprofen up to 2400 mg; With at least 128 participants, the study had a 92% power to establish that etoricoxib is noninferior to ibuprofen (null hypothesis). The power and sample size were based on the following assumptions: 1) an approximately 15% protocol violation rate, 2) a noninferiority margin of -3.7 units (etoricoxib minus ibuprofen), and 3) an intrapatient standard deviation of 8 units; Test type: Non-Inferiority or Equivalence — The noninferiority margin is -3.7 units; p = 0.043, ANOVA — A priori threshold for statistical significance = <0.025 (one-sided); Adjusted for treatment, period, sequence, patient (sequence), and baseline pain intensity (moderate or severe); Difference in LS Means = 0.89, 95% CI 2-sided [0.03 to 1.76]

2. Secondary Outcome: Sum of Pain Intensity Difference Scores Over the 6-Hour Time Period (SPID6)
Description: The Pain Intensity Difference (PID) score is the difference between the baseline pain intensity (PI) score and the PI score recorded at each time point post initial dose, as calculated by subtracting the pain intensity at each of the subsequent time points from the baseline pain intensity score; therefore, it is on a -1 to 3 scale, with a large value representing a greater treatment effect. SPID6 is derived by multiplying the PID score at each time point by the duration (in hours) since the preceding time point, and summing these weighted values up to 6 hours and it is on a scale of -6 to 18.
Time Frame: Baseline and 0.5, 1, 1.5, 2, 3, 4, 5 and 6 hours
Population: The population consisted of all participants that received at least one dose of study treatment, had at least one SPID6 observation up to 6 hours post initial dose of study medication, and had a baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Etoricoxib 120 mg | Ibuprofen up to 2400 mg
Number analyzed (Participants) | 130 | 130
Score on a Scale | 9.48 (0.58) | 9.27 (0.58)
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Ibuprofen up to 2400 mg; Test type: Superiority or Other; p = 0.768, ANOVA — A nominal threshold for statistical significance = <0.05; Adjusted for treatment, period, sequence, patient (sequence), and baseline pain intensity (moderate or severe); Difference in LS Means = 0.20, 95% CI 2-sided [-1.16 to 1.57]

3. Secondary Outcome: Mean Participant Global Evaluation of Pain at 6 Hours After the Initial Dose (GLOBAL6)
Description: The GLOBAL6 was recorded by the participant at 6 hours (or at the time of rescue medication use) after taking the first dose of study medication. The GLOBAL6 uses a pain relief scale of 0 to 4, where 0 = poor pain relief, 1 = fair pain relief, 2 = good pain relief, 3 = very good pain relief, and 4 = excellent pain relief.
Time Frame: 6 hours
Population: The population consisted of all participants that received at least one dose of study treatment and had a GLOBAL6 observation at 6 hours post initial dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Etoricoxib 120 mg | Ibuprofen up to 2400 mg
Number analyzed (Participants) | 129 | 129
Score on a Scale | 2.50 (0.08) | 2.24 (0.08)
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Ibuprofen up to 2400 mg; Test type: Superiority or Other; p = 0.007, ANOVA — A nominal threshold for statistical significance = <0.05; Adjusted for treatment, period, sequence, patient (sequence), and baseline pain intensity (moderate or severe); Difference in LS Means = 0.26, 95% CI 2-sided [0.07 to 0.45]

4. Secondary Outcome: Mean Participant Global Evaluation of Pain at 24 Hours After the Initial Dose (GLOBAL24)
Description: The GLOBAL24 was recorded by the participant at 24 hours (or at the time of rescue medication use) after taking the first dose of study medication. The GLOBAL24 uses a pain relief scale of 0 to 4, where 0 = poor pain relief, 1 = fair pain relief, 2 = good pain relief, 3 = very good pain relief, and 4 = excellent pain relief.
Time Frame: 24 hours
Population: The population consisted of all participants that received at least one dose of study treatment had a GLOBAL24 observation at 24 hours post initial dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Etoricoxib 120 mg | Ibuprofen up to 2400 mg
Number analyzed (Participants) | 129 | 129
Score on a Scale | 2.65 (0.08) | 2.29 (0.08)
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Ibuprofen up to 2400 mg; Test type: Superiority or Other; p < 0.001, ANOVA — A nominal threshold for statistical significance = <0.05; Adjusted for treatment, period, sequence, patient (sequence), and baseline pain intensity (moderate or severe); Difference in LS Means = 0.36, 95% CI 2-sided [0.17 to 0.54]

5. Secondary Outcome: Mean Time to >=1 Unit Improvement From Baseline in Pain Intensity During the 6 Hours After the Initial Dose
Description: The time to a change from baseline in pain intensity score of >=1 unit on the pain intensity scale was calculated. The pain intensity scale rates participant pain on a scale of -1 to 3, with larger values associated with greater treatment effect.
Time Frame: Baseline and 6 hours
Population: The population consisted of all participants that received at least one dose of study treatment, had an observation at 6 hours post initial dose of study medication, and had a baseline measurement.
Measure: Mean (95% Confidence Interval); unit: Hours
Arm/Group | Etoricoxib 120 mg | Ibuprofen up to 2400 mg
Number analyzed (Participants) | 130 | 130
Hours | 1.0 [1.0 to 1.5] | 1.5 [1.0 to 1.5]
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Ibuprofen up to 2400 mg; Test type: Superiority or Other; p = 0.371, Regression, Cox — A priori threshold for statistical significance = <0.05; Adjusted for treatment, period, and baseline pain intensity; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.70 to 1.14]

6. Secondary Outcome: Peak Pain Intensity Difference (PID) During the 6 Hours After the Initial Dose
Description: Peak PID during the 6 hours post initial dose is defined as the maximum PID score recorded during first 6 hours after the initial dose of study medication. PID is evaluated on a scale of -1 to 3, with larger values representing a greater treatment effect.
Time Frame: Baseline and 0.5, 1, 1.5, 2, 3, 4, 5 and 6 hours
Population: The population consisted of all participants that received at least one dose of study treatment and had a PID observation at up to 6 hours post initial dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Etoricoxib 120 mg | Ibuprofen up to 2400 mg
Number analyzed (Participants) | 130 | 130
Score on a Scale | 2.2 (0.4) | 2.1 (0.4)
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Ibuprofen up to 2400 mg; Test type: Superiority or Other; p = 0.051, ANOVA — A priori threshold for statistical significance = <0.05; Adjusted for treatment, period, sequence, patient (sequence), and baseline pain intensity (moderate or severe); Difference in LS Means = 0.10, 95% CI 2-sided [-0.00 to 0.20]

7. Secondary Outcome: Peak Pain Relief (Peak PR) During the 6 Hours After the Initial Dose
Description: Peak PR during the 6 hours post initial dose is defined as the maximum PR score
  recorded during the first 6 hours after the initial dose of study medication. PR is recorded on a scale of 0 to 4, with 0 = no pain relief, 1 = little pain relief, 2 = some pain relief, 3 = a lot of pain relief, and 4 = complete pain relief.
Time Frame: Up to 6 hours
Population: The population consisted of all participants that received at least one dose of study treatment and had at least one Peak PR observation up to 6 hours post initial dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Etoricoxib 120 mg | Ibuprofen up to 2400 mg
Number analyzed (Participants) | 130 | 130
Score on a Scale | 3.70 (0.06) | 3.52 (0.06)
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Ibuprofen up to 2400 mg; Test type: Superiority or Other; p = 0.019, ANOVA — A priori threshold for statistical significance = <0.05; Adjusted for treatment, period, sequence, patient (sequence), and baseline pain intensity (moderate or severe); Mean Difference in LS Means = 0.17, 95% CI 2-sided [0.03 to 0.32]

8. Secondary Outcome: Number of Participants Using Rescue Medication 24 Hours After the Initial Dose
Description: Acetaminophen 250 mg, isopropylantipyrine 150 mg and anhydrous caffeine 50 mg (Saridon) was provided to each participant as rescue medication. Participants were permitted to take 2 tablets at a time and up to 3 doses within 24 hours of dosing of study drug for rescue purposes.
Time Frame: 24 Hours
Population: Due to the low number of participants requiring rescue medication use, the time to rescue medication use was not calculated.
Measure: Number; unit: Participants
Arm/Group | Etoricoxib 120 mg | Ibuprofen up to 2400 mg
Number analyzed (Participants) | 130 | 130
Participants | 1 | 4

9. Secondary Outcome: PID at Up to 12 Hours Following the Initial Dose
Description: PID during the 12 hours following the initial dose is defined as the maximum PID score recorded during first 12 hours after the initial dose of study medication. PID is evaluated on a scale from 0 to 3, with 0 = no pain, 1 = slight pain, 2 = moderate pain, and 3 = severe pain.
Time Frame: Baseline and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8 and 12 hours
Population: The population consisted of all participants that received at least one dose of study treatment and had at least one PID observation at up to 12 hours post initial dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Etoricoxib 120 mg | Ibuprofen up to 2400 mg
Number analyzed (Participants) | 130 | 129
Score on a Scale | 2.28 (0.04) | 2.07 (0.04)
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Ibuprofen up to 2400 mg; Test type: Superiority or Other; p < 0.001, ANOVA — A priori threshold for statistical significance = <0.05; Adjusted for treatment, period, sequence, patient (sequence), and baseline pain intensity (moderate or severe); Difference in LS Means = 0.21, 95% CI 2-sided [0.10 to 0.31]

10. Secondary Outcome: PR at Up to 12 Hours Following the Initial Dose
Description: PR during the 12 hours following the initial dose is defined as the maximum PR score recorded during the first 12 hours after the initial dose of study medication. PR is evaluated on a scale of 0 to 4, with 0 = no pain relief, 1= a little pain relief, 2 = some pain relief, 3 = a lot of pain relief, and 4 = complete pain relief.
Time Frame: Up to 12 hours
Population: The population consisted of all participants that received at least one dose of study treatment and had at least one PR observation up to 12 hours post initial dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Etoricoxib 120 mg | Ibuprofen up to 2400 mg
Number analyzed (Participants) | 130 | 129
Score on a Scale | 3.73 (0.07) | 3.45 (0.07)
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Ibuprofen up to 2400 mg; Test type: Superiority or Other; p = 0.002, ANOVA — A priori threshold for statistical significance = <0.05; Adjusted for treatment, period, sequence, patient (sequence), and baseline pain intensity (moderate or severe); Difference in LS Means = 0.28, 95% CI 2-sided [0.10 to 0.45]

11. Secondary Outcome: PID at Up to 24 Hours Following the Initial Dose
Description: PID during the 24 hours following the initial dose is defined as the maximum PID score recorded during first 24 hours after the initial dose of study medication. PID is evaluated on a scale from 0 to 3, with 0 = no pain, 1 = slight pain, 2 = moderate pain, and 3 = severe pain.
Time Frame: Baseline and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 20 and 24 hours
Population: The population consisted of all participants that received at least one dose of study treatment and had at least one PID observation up to 24 hours post initial dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Etoricoxib 120 mg | Ibuprofen up to 2400 mg
Number analyzed (Participants) | 130 | 130
Score on a Scale | 2.36 (0.04) | 2.25 (0.04)
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Ibuprofen up to 2400 mg; Test type: Superiority or Other; p = 0.011, ANOVA — A priori threshold for statistical significance = <0.05; Adjusted for treatment, period, sequence, patient (sequence), and baseline pain intensity (moderate or severe); Difference in LS Means = 0.11, 95% CI 2-sided [0.03 to 0.20]

12. Secondary Outcome: PR at Up to 24 Hours Following the Initial Dose
Description: PR during the 24 hours following the initial dose is defined as the maximum PR score recorded during the first 24 hours after the initial dose of study medication. PR is evaluated on a scale of 0 to 4, with 0 = no pain relief, 1= a little pain relief, 2 = some pain relief, 3 = a lot of pain relief, and 4 = complete pain relief.
Time Frame: Up to 24 hours
Population: The population consisted of all participants that received at least one dose of study treatment and had at least one PR observation at up to 24 hours post initial dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Etoricoxib 120 mg | Ibuprofen up to 2400 mg
Number analyzed (Participants) | 130 | 130
Score on a Scale | 3.88 (0.07) | 3.62 (0.07)
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Ibuprofen up to 2400 mg; Test type: Superiority or Other; p = 0.004, ANOVA — A priori threshold for statistical significance = <0.05; Adjusted for treatment, period, sequence, patient (sequence), and baseline pain intensity (moderate or severe); Difference in LS Means = 0.26, 95% CI 2-sided [0.08 to 0.44]

13. Secondary Outcome: Number of Participants With a Global Evaluation of Study Medication of Good, Very Good, or Excellent at 6 Hours After the Initial Dose
Description: At 6 hours following the initial dose. participants were asked to rate their perception of pain control as poor, fair, good, very good, or excellent. The number of participants that reported good, very good, or excellent pain control at 6 hours post initial dose were summed.
Time Frame: 6 hours
Population: The population consisted of all participants that received at least one dose of study treatment and completed the assessment at 6 hours post initial dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Etoricoxib 120 mg | Ibuprofen up to 2400 mg
Number analyzed (Participants) | 129 | 129
Participants | 111 | 103
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Ibuprofen up to 2400 mg; Test type: Superiority or Other; p = 0.112, Regression, Logistic — A priori threshold for statistical significance = <0.05; Adjusted for treatment, period, and baseline pain intensity; Odds Ratio (OR) = 1.60, 95% CI 2-sided [0.90 to 2.87]

14. Secondary Outcome: Number of Participants With a Global Evaluation of Study Medication of Good, Very Good, or Excellent at 24 Hours After the Initial Dose
Description: At 24 hours following the initial dose of study medication, participants were asked to rate their perception of pain control as poor, fair, good, very good, or excellent. The number of participants that reported good, very good, or excellent pain control at 24 hours post initial dose were summed.
Time Frame: 24 Hours
Population: The population consisted of all participants that received at least one dose of study treatment and completed the assessment at 24 hours post initial dose of study medication
Measure: Number; unit: Participants
Arm/Group | Etoricoxib 120 mg | Ibuprofen up to 2400 mg
Number analyzed (Participants) | 129 | 129
Participants | 113 | 101
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Ibuprofen up to 2400 mg; Test type: Superiority or Other; p = 0.019, Regression, Logistic — A priori threshold for statistical significance = <0.05; Adjusted for treatment, period, and baseline pain intensity; Odds Ratio (OR) = 1.97, 95% CI 2-sided [1.12 to 3.45]

ADVERSE EVENTS:
Time Frame: From the time of the initial (first) dose of study medication up to 14 days after last dose of study medication.
Description: The safety population consisted of all randomized participants who received at least 1 dose of study treatment in at least 1 treatment cycle. For each treatment cycle, participants were to be included in the study treatment they actually received for the analysis of safety data.
Groups:
- Etoricoxib 120 mg / Ibuprofen up to 2400 mg/Daily: Etoricoxib 120 mg tablet given orally for one dose in menstrual cycle 1. In menstrual cycle 2, ibuprofen was administered at a dose of 600 mg every 4 hours as needed up to 2400 mg/day.
- Ibuprofen up to 2400 mg / Etoricoxib 120 mg: Ibuprofen 600 mg given orally up to four times a day as needed, for a maximum of 2400 mg/day in menstrual cycle 1. In menstrual cycle 2, etoricoxib was administered at a dose of 120 mg daily.
Arm/Group | Etoricoxib 120 mg / Ibuprofen up to 2400 mg/Daily | Ibuprofen up to 2400 mg / Etoricoxib 120 mg
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/70
Other Adverse Events (participants affected / at risk) | 0/69 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. The sponsor review can be expedited to meet publication timelines.